CLINICAL TRIAL: NCT02647203
Title: Non-invasive Therapy With Fluoridated Toothpastes for Root Caries in Independently-living Older Adults
Brief Title: Non-invasive Treatment of Root Caries in Older Adults
Acronym: MIT-RCTalca
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Talca (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Rodrigo A. Giacaman, DDS, PhD, Associate Professor, University of Talca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NI-RC PIEI-ES; 1140623 (Other Grant/Funding Number: Fondecyt - Conicyt Chile)
Record Dates: First submitted 2015-12-07; First posted 2016-01-06 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2020-12

CONDITIONS: Root Caries
Keywords: Fluoride toothpaste; Root caries; Randomized clinical trial
MeSH Terms: conditions — Root Caries | interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Fluoride Toothpaste (Experimental): 5,000 ppm fluoridated toothpaste, high concentration. Self-administered fluoridated dentifrices. By the elderly subjects, twice per day Drug (including placebo)
  Interventions: Drug: Self-administered fluoridated dentifrices
- Standard Fluoride Toothpaste (Active Comparator): 1,450 ppm fluoridated toothpaste, low concentration. Self-administered fluoridated dentifrices. By the elderly subjects, twice per day Drug (including placebo)
  Interventions: Drug: Self-administered fluoridated dentifrices

INTERVENTIONS:
Drug: Self-administered fluoridated dentifrices — Elderly participants will be instructed to self administer toothpastes, twice per day. Toothpastes will be provided.
  Other Names: Toothbrushing with high and standard fluoride dentifrices

SUMMARY:
This study aims to test the effectiveness in reducing or arresting root caries lesion in community-dwelling elderly subjects by using high fluoridated toothpaste. A double blinded RCT will be conducted with two arms; 5000 ppm F and 1450 ppm F toothpaste. Dentifrices will be delivered to the participants in a blind format and they will be instructed to brush twice per day.

Follow-up will be carries out every 6 months for two years to assess:

* Root caries incidence.
* Lesion arresting
* Changes in salivary flow
* Microbiology pattern shift
* Variations in oral health- related quality of life by OHIP-14 Sp

DETAILED DESCRIPTION:
Background. Caries of the root surface (root caries) is the most prevalent type of dental caries in older adults with a reportedly worrisome trend to increase, as more teeth are being retained. Dental caries is the leading causes of tooth loss among older adults. Fluoride has been successfully used in preventive programs for root caries. In addition to preventing root caries, fluoride-based therapies may be used to treat lesions. This approach is known as non-invasive treatment. Fluoride seems to arrest and promote remineralization of the lesions. Indeed, recent studies appear to indicate that, higher fluoride concentrations are more effective to prevent and to treat the disease. Dentifrices with high concentrations of fluoride appear to be the most rational approach to prevent and treat root caries. To the chemical effect of fluoride, toothbrushing adds mechanical removal of the dental biofilm. High concentration fluoride varnishes have also been proposed as effective in treating carious lesions. Whether dentifrices, varnishes or the combined use of varnish and fluoridated toothpaste result more effective is a matter of controversy and it needs to be elucidated. Non-invasive treatment avoids the complications inherent to treating frail people in a dental setting, decrease costs and importantly, allows increased coverage, as these therapies may be delivered by non-dentist personnel. Although the appealing idea of non-invasive treatment of root caries in older adults, evidence is still limited and more research appears necessary to both, confirm clinical success and elucidate the mechanisms involved in lesion arrestment.

Aim. To determine the effectiveness of non-invasive therapies for root caries and their impact in the quality of life of older adults.

Methodology. A double blind randomized controlled trial (RCT) on independently-living older adults aged sixty or more years is proposed. Subjects will undergo clinical and microbiological examination when recruited (baseline) with a six-month follow-up regime until completion of two years. To participate, subjects will have to have at least five teeth with exposed root surfaces and one carious lesion. Sample size was calculated and a sample of two-hundred and eighty-eight older adults is necessary, randomized into two study arms;

Group 1: toothpaste 1.450 ppm F-

Group 2: toothpaste 5.000 ppm F-

Dependent variables. Root caries incidence and activity, cariogenic bacteria and oral health-related quality of life will be assessed upon completion of the study and compared with baseline scores.

Expected results. Based on some previous data available, it is expected that a non-invasive therapy for root caries based on low-fluoride concentration will be less effective than high fluoride therapies in inactivating root caries lesions. These results may be used in novel therapeutic programs at the community level, as well as in private practice. Furthermore, these studies will shed light on potential mechanisms associated with non-invasive treatment of root caries, from a microbiology stand point. Since a non-invasive approach decreases costs and increases coverage of dental care for older adults, these results may contribute to increase access to care for the usually vulnerable population of older adults.

ELIGIBILITY:
Inclusion Criteria:

* 60 + years old
* community-dwelling
* living in a community with fluoridated water
* had five or more of their own teeth
* with ≥ 1 root caries lesion

Exclusion Criteria:

* cognitive impairment
* alcoholism

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo A Giacaman, DDS, PhD, Principal Investigator — University of Talca
Locations (1):
- Faculty of Health Sciences, Talca, No State, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ekstrand K, Martignon S, Holm-Pedersen P. Development and evaluation of two root caries controlling programmes for home-based frail people older than 75 years. Gerodontology. 2008 Jun;25(2):67-75. doi: 10.1111/j.1741-2358.2007.00200.x. Epub 2008 Jan 13. PMID 18194330
- [Background] Ekstrand KR, Poulsen JE, Hede B, Twetman S, Qvist V, Ellwood RP. A randomized clinical trial of the anti-caries efficacy of 5,000 compared to 1,450 ppm fluoridated toothpaste on root caries lesions in elderly disabled nursing home residents. Caries Res. 2013;47(5):391-8. doi: 10.1159/000348581. Epub 2013 Apr 9. PMID 23594784
- [Background] Gluzman R, Katz RV, Frey BJ, McGowan R. Prevention of root caries: a literature review of primary and secondary preventive agents. Spec Care Dentist. 2013 May-Jun;33(3):133-40. doi: 10.1111/j.1754-4505.2012.00318.x. Epub 2012 Dec 10. PMID 23600985
- [Background] Griffin SO, Griffin PM, Swann JL, Zlobin N. Estimating rates of new root caries in older adults. J Dent Res. 2004 Aug;83(8):634-8. doi: 10.1177/154405910408300810. PMID 15271973
- [Background] Griffin SO, Regnier E, Griffin PM, Huntley V. Effectiveness of fluoride in preventing caries in adults. J Dent Res. 2007 May;86(5):410-5. doi: 10.1177/154405910708600504. PMID 17452559
- [Background] Holmgren C, Gaucher C, Decerle N, Domejean S. Minimal intervention dentistry II: part 3. Management of non-cavitated (initial) occlusal caries lesions--non-invasive approaches through remineralisation and therapeutic sealants. Br Dent J. 2014 Mar;216(5):237-43. doi: 10.1038/sj.bdj.2014.147. PMID 24603245
- [Background] Ritter AV, Shugars DA, Bader JD. Root caries risk indicators: a systematic review of risk models. Community Dent Oral Epidemiol. 2010 Oct;38(5):383-97. doi: 10.1111/j.1600-0528.2010.00551.x. PMID 20545716
- [Background] Walls AW, Meurman JH. Approaches to caries prevention and therapy in the elderly. Adv Dent Res. 2012 Sep;24(2):36-40. doi: 10.1177/0022034512453590. PMID 22899677
- [Result] Leon S, Bravo-Cavicchioli D, Correa-Beltran G, Giacaman RA. Validation of the Spanish version of the Oral Health Impact Profile (OHIP-14Sp) in elderly Chileans. BMC Oral Health. 2014 Aug 4;14:95. doi: 10.1186/1472-6831-14-95. PMID 25091189
- [Derived] Leon S, Gonzalez K, Hugo FN, Gambetta-Tessini K, Giacaman RA. High fluoride dentifrice for preventing and arresting root caries in community-dwelling older adults: A randomized controlled clinical trial. J Dent. 2019 Jul;86:110-117. doi: 10.1016/j.jdent.2019.06.002. Epub 2019 Jun 6. PMID 31176788
- See also: CEPAL (2013). Observatorio demográfico 2012. Proyecciones de población — https://repositorio.cepal.org/bitstream/handle/11362/7118/1/S2012922_mu.pdf
- See also: ONS (2013). Statistical bulletin: National Population Projections, 2012-based Statistical Bulletin — http://www.ons.gov.uk/ons/rel/npp/national-population-projections/2012-based-projections/stb-2012-based-npp-principal-and-key-variants.html

RESULTS

PARTICIPANT FLOW:
Period: 12 Month Follow-up
Arm/Group | High Fluoride Toothpaste | Standard Fluoride Toothpaste
Started | 173 | 172
Completed | 148 | 149
Not Completed | 25 | 23
Period: 24 Month Follow-up
Arm/Group | High Fluoride Toothpaste | Standard Fluoride Toothpaste
Started | 148 | 149
Completed | 142 | 138
Not Completed | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Fluoride Toothpaste | Standard Fluoride Toothpaste | Total
Number analyzed (Participants) | 173 | 172 | 345
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 173 | 172 | 345
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 127 | 258
  Male | 42 | 45 | 87
Socioeconomic status [Count of Participants; unit: Participants]
  Upper | 64 | 60 | 124
  Lower | 109 | 112 | 221
Education [Count of Participants; unit: Participants]
  Less or equal than 8 years | 42 | 51 | 93
  9 - 12 years | 70 | 57 | 127
  More than 12 years | 61 | 64 | 125

OUTCOME MEASURES:

1. Primary Outcome: Root Caries Activity
Description: Using Nyvad's criteria for root caries lesions, activity will be assessed by a visual-tactile method.
Time Frame: After 2 years of follow up
Population: Independently-living older adults
Measure: Mean (Standard Deviation); unit: Percentage of active lesions (2-years)
Arm/Group | High Fluoride Toothpaste | Standard Fluoride Toothpaste
Number analyzed (Participants) | 142 | 138
Percentage of active lesions (2-years) | 3.72 (12.32) | 40.52 (23.30)

2. Secondary Outcome: Oral Health Related Quality of Life, Measured by the Oral Health Impact Profile (OHIP-14 Sp)
Description: The impact on the quality of life of the therapy will be explored using the OHIP-14 Sp, validated by our group. In a scale ranging from 0 to 56 points, with 0-14 being good Oral Health-related quality of life and 15-56 poor Oral Health-related quality of life.
Time Frame: Data registered at 2 years of follow-up
Population: Independently-living older adults
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Fluoride Toothpaste | Standard Fluoride Toothpaste
Number analyzed (Participants) | 143 | 137
score on a scale | 10.71 (9.56) | 11.28 (9.25)

3. Secondary Outcome: Salivary Flow
Description: Unstimulated Salivary Flow, defined as Normal or Low Important: This outcome measure was originally considered. However, due to logistic issues, we did not assess it and no data is available.
Time Frame: Baseline and 2-year follow up
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: 2 years
Description: Burning feeling, irritation or feeling the mouth uncomfortably are the only potential adverse effects, due to the dentifrices used.
  All-Cause Mortality was monitored/assessed
Arm/Group | High Fluoride Toothpaste | Standard Fluoride Toothpaste
All-Cause Mortality (participants affected / at risk) | 0/142 | 0/138
Serious Adverse Events (participants affected / at risk) | 0/142 | 0/138
Other Adverse Events (participants affected / at risk) | 0/142 | 0/138

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No